CLINICAL TRIAL: NCT04248387
Title: A Clinical Study on the Efficacy and Safety of Toripalimab in the Neoadjuvant Treatment of BRAF V600 Wild Type Resectable Stage III / IV Malignant Melanoma
Brief Title: Toripalimab in the Neoadjuvant Treatment of BRAF V600 Wild Type Melanoma
Acronym: FU-Name-T001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yong Chen, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB1906203-3
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Melanoma Stage IIIB-IV
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab group (Experimental): The subjects in this group receive intravenous drip infusion of Toripalimab at a dose of 3 mg / kg once every 2 weeks for a total of two cycles
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Toripalimab, intravenous drip infusion, a dose of 3 mg / kg once every 2 weeks for a total of two cycles
  Other Names: JS001

SUMMARY:
In view of the fact that neoadjuvant therapy for malignant melanoma is in the exploratory stage, and the current data on neoadjuvant immunology are mainly from European and American populations, it is necessary to carry out clinical trials in the status of neoadjuvant immunotherapy for patients with melanoma in China. Toripalimab has been extensively studied in the field of malignant melanoma, and its effectiveness and safety have been proven. Therefore, the investigators initiated a single-arm exploratory study to investigate the efficacy and safety of Toripalimab in neoadjuvant treatment of patients with BRAF V600 wild-type malignant melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can undergo surgery after discussion by three surgeons with a deputy senior title or higher
* Patients with stage III or oligometastasis stage IV malignant melanoma confirmed by histopathology or cytology. Stage III is defined as at least one clinically accessible lymph node metastasis; oligometastasis stage IV is defined as less than 4 metastases and the site of metastasis excludes bone metastases, brain metastases, or other metastases that cannot be completely surgically treated.
* BRAF V600 wild type
* Age ≥ 18 years old
* ECOG score is 0-1, with an estimated overall survival of more than 1 year
* The function of main organs and bone marrow is basically normal:

  1. Blood routine: WBC ≥ 3500 / mm3 (3.5 * 109 / L); Neutrophil count (ANC) ≥ 180 / mm3 (1.8 * 109 / L); Platelet count ≥ 125000 / mm3 (125 * 109 / L); Hemoglobin: male ≥ 13g / dl (130g / L); female ≥ 11.5g/dl (115g / L);
  2. Blood biochemistry: Total bilirubin ≤ 1.5 * ULN (total bilirubin of Gilbert syndrome <3.0mg / dL); Aspartate aminotransferase (AST / SGOT), alanine aminotransferase (ALT / SGPT) and alkaline phosphatase ≤ 2.5 * ULN; Creatinine ≤1.5 * normal upper limit (ULN);
  3. Coagulation function: The international standard ratio (INR) is less than 1.5 (or the INR value is 2-3 when patients take farwarin stably for a long time), and prothrombin time (PT) is less than 1.5 * ULN;
  4. Lung function test: Lung diffusion (DLCO) ≥ 70% predicted OR; DLCO <70% but ≥ 55%, and the maximum oxygen uptake (VO2 max) ≥ 10L / min / kg (by cardiopulmonary assessment) or 6 minutes walking test ≥ 500 meters; Patients with DLCO <55% were not included in this study; Pulse oximetry during rest and walking ≥ 92%;
  5. Heart function test: Baseline ECG showed no prolonged PR interval or atrioventricular block;
* Women should agree to use contraceptive measures (such as intrauterine device (IUD), contraceptive or condom) during the study and within 6 months after the end of the study; women should be negative in serum or urine pregnancy test within 7 days before the study and must be non lactating; men should agree to use contraceptive measures during the study and within 6 months after the end of the study.
* Patients voluntarily joined the study, signed informed consent, and had good compliance and were able to be followed up by the trial staff.

Exclusion Criteria:

* A previous history of activity or history of any autoimmune disease (including any history of inflammatory bowel disease), or a history of syndrome requiring treatment with systemic steroids or immunosuppressive drugs (except vitiligo patients);
* Use vaccines against infectious diseases (such as influenza, varicella, etc.) within 4 weeks (28 days) after the start of the study treatment;
* Active systemic infection requiring treatment, positive detection of hepatitis B surface antigen or hepatitis C ribonucleic acid (RNA);
* A known positive medical history or positive test result for human immunodeficiency virus or acquired immunodeficiency syndrome (AIDS);
* Patients with any serious and / or uncontrollable diseases, such as unstable angina, symptomatic congestive heart failure, myocardial infarction within 6 months before randomization, serious uncontrollable arrhythmia; patients with poor blood pressure control (systolic pressure > 140 mmHg, diastolic pressure > 90 mmHg); active or uncontrollable serious infection; liver diseases such as cirrhosis , decompensated liver disease, chronic active hepatitis; poor control of diabetes mellitus (FBG > 10mmol / L); routine urine test indicated that urine protein was ≥ + +, and confirmed that 24-hour urine protein quantity was > 1.0g;
* A history of psychotropic substance abuse who are unable to quit or have a mental disorder;
* Have been previously exposed to any anti-tumor treatment, including but not limited to chemotherapy, radiotherapy, immunotherapy (such as anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-CTLA-4 antibody or any other antibody targeting T-cell co regulatory pathway), etc.; are currently using tumor related treatment or online anti-cancer drugs; are currently using anticoagulants; have received large-scale surgical treatment in the past 3 weeks;
* Previously had malignant tumors and did not achieve complete remission at least 2 years before the start of the study without other treatments (except skin basal cell carcinoma or cervical carcinoma in situ)；
* A history of previous interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis, symptomatic interstitial lung disease, or chest CT scans found any evidence of active pneumonia within 4 weeks before the first study medication;
* Immunosuppressive drugs were used within 2 weeks before the first study drug treatment, excluding local glucocorticoids or prednisone with systemic glucocorticoids no more than 10 mg / day or other glucocorticoids of equivalent dose;
* Pregnant or lactating women;
* Prisoners who have been illegally imprisoned or detained for non-mental or physical (such as infectious) diseases;
* Patients with a bleeding tendency (such as active peptic ulcer) or treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogs;
* A history of allergy to the ingredients of the study drug;
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of patients or affect patients to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate | Within one week after operation
  Pathologic complete response rate

SECONDARY OUTCOMES:
EFS rate | One year after the first intravenous drip
  Event-free survival rate
ORR | One year after the first intravenous drip
  Objective response rate
OS | Three years after the first intravenous drip
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.